CLINICAL TRIAL: NCT05971615
Title: Evaluate the Relevance of the Use of Peripheral Venous Blood Gases for the Care of Patients in the S.A.U.V (Vital Emergency Rooms) of the CHU de Caen
Acronym: GDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-076
Record Dates: First submitted 2023-05-23; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peripheral Venous Blood Gases (Other)
  Interventions: Other: peripheral venous blood gases

INTERVENTIONS:
Other: peripheral venous blood gases — peripheral venous blood gases

SUMMARY:
concordance between the lactate values on peripheral venous and arterial blood gases in all patients receiving an arterial sample on their arrival in the S.A.U.V.

ELIGIBILITY:
Inclusion Criteria:

* one of this condition in emergency unit :

  1. acute respiratory distress
  2. a suspicion of an acid-base disorder
  3. a state of shock
  4. Pathologies requiring monitoring of the respiratory system
  5. Patient under NIV
  6. Poisoning
  7. Coma with a Glasgow score < or equal to 8

Exclusion Criteria:

* Patient presenting another pathology supported in SAUV not requiring the realization of arterial blood gases
* Patient aged < 18 years
* Pregnant or breastfeeding woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
lactates on peripheral venous and arterial blood gases | baseline
  mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No